CLINICAL TRIAL: NCT02354690
Title: T-cell Therapy in Combination With Vemurafenib for Patients With BRAF Mutated Metastatic Melanoma
Brief Title: Vemurafenib and TIL Therapy for Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Professor, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM1414
Record Dates: First submitted 2015-01-26; First posted 2015-02-03 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; Cyclophosphamide; fludarabine; Adoptive Transfer; Immunotherapy, Adoptive; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): 7 days before tumor harvest, patients will begin taking vemurafenib until admission for lymphodepleting chemotherapy regimen of cyclophosphamide and fludarabine, followed by TIL infusion and interleukin-2.
  Interventions: Drug: Vemurafenib; Drug: Lymphodepleting chemotherapy; Drug: TIL infusion; Drug: Interleukin-2

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib is used to treat patients with BRAF mutated metastatic melanoma. Patients will start treatment in a dose of 960 BID 7 days before tumor harvest and ends at the day of admission (day -8).
  Other Names: Zelboraf; BRAF inhibitor
Drug: Lymphodepleting chemotherapy — First patients undergo lymphodepleting chemotherapy regimen consisting of cyclophosphamide 60 mg/kg for 2 days and fludarabine 25 mg/m2 for 5 days (constitutes day -7 to -1 of admission).
  Other Names: cyclophosphamide; fludarabine
Drug: TIL infusion — 7 days after start of vemurafenib treatment, patients undergo surgery to removal of a tumor in order to isolate, activate and expand tumor infiltrating lymphocytes (TIL) to high numbers. In vitro preparation usually takes 4-6 weeks using the young TIL method.
  On day 0 patients receive an infusion of TIL (1x10e9-2x10e11 cells).
  Other Names: Adoptive cell transfer; T cell therapy
Drug: Interleukin-2 — After infusion of TILs, patients will receive interleukin-2 infusions according to the decrescendo regimen (18 MIU/m2 for 6 hours, 18 MIU/m2 for 12 hours, 18 MIU/m2 for 24 hours followed by 4,5 MIU/m2 for another 3 x 24 hours)
  Other Names: IL-2

SUMMARY:
Background:

Adoptive T cell therapy with tumor infiltrating lymphocytes (TILs) has been reported to induce durable clinical responses in patients with metastatic melanoma. From patients own tumor material T cells are extracted, expanded and activated in vitro in a 4-6 weeks culture period. Before TIL infusion patients are preconditioned with a lymphodepleting chemotherapeutic regimen. After TIL infusion, patients are treated with IL-2 to support T cell activation and expansion in vivo.

The BRAF inhibitor is an approved treatment of metastatic melanoma and functions by selectively inhibiting the BRAF mutated enzyme, consequently halting the proliferation of tumor cells. Furthermore, in vitro tests have shown that vemurafenib has immunomodulatory effects that are hypothesized to synergize with TIL therapy, which has been confirmed in animal studies.

Objectives:

* To evaluate safety and feasibility when combining vemurafenib and ACT with TILs.
* To evaluate treatment related immune responses
* To evaluate clinical efficacy

Design:

* Patients will be screened with a physical exam, medical history, blood samples and ECG.
* Patients will start vemurafenib 960 mg BID and will continue during TIL preparation.
* 7 days after start of vemurafenib, patients will undergo surgery to harvest tumor material for TIL production.
* Patient stops vemurafenib and is admitted day -8 in order to undergo lymphodepleting chemotherapy with cyclophosphamide and fludara starting day -7.
* On day 0 patients receive TIL infusion and shortly after starts IL-2 infusion continually following the decrescendo regimen.
* The patients will followed until progression or up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable stage III or stage IV metastatic melanoma.
* Metastasis available for surgical resection (about 2 cm3) and residual measureable disease after resection.
* Pathologically verified BRAF mutation.
* ECOG performance status 0-1.
* Life expectancy ≥ 3 months.
* No significant toxicity (CTC ≤ 1) from prior treatments.
* Adequate renal, hepatic and hematologic function.
* Women of childbearing potential (WOCBP) and men in a sexual relationship with a WOCBP must be using an effective method of contraception during treatment and for at least 6 months after completion of treatment.
* Able to comprehend the information given and willing to sign informed consent.

Exclusion Criteria:

* Other malignancies, unless followed for ≥ 5 years with no sign of disease, except squamous cell carcinoma or adequately treated carcinoma in situ colli uteri.
* Cerebral metastasis. Patients with previously treated CNS metastasis can participate if surgically removed or treated with stereotactic radiotherapy if stable > 28 days after treatment measured by MRI. Patients with asymptomatic and untreated CNS metastasis can participate based on investigators evaluation.
* Patients with ocular melanoma.
* Previous treatment with a BRAF inhibitor.
* Severe allergies, history of anaphylaxis or known allergies to drugs administered.
* Serious medical or psychiatric comorbidity.
* QTc ≥ 450 ms.
* Clearance < 70 ml/min.
* Acute or chronic infection with e.g. HIV, hepatitis, tuberculosis
* Active autoimmune disease.
* Pregnant og nursing women.
* Need for immunosuppressive treatment, e.g. corticosteroids or methotrexate.
* Concomitant treatment with other experimental drugs.
* Patients with uncontrolled hypercalcemia
* More than four weeks must have elapsed since any prior systemic therapy at the time of treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Prof., MD, Study Director — Department of Oncology, Copenhagen University Hospital, Herlev, Herlev Ringvej 75, DK-2730 Herlev, Denmark; Troels Holz Borch, MD, Principal Investigator — Department of Oncology, Copenhagen University Hospital, Herlev, Herlev Ringvej 75, DK-2730 Herlev, Denmark
Locations (1):
- Center for Cancer Immune Therapy, Dept. of Haematology/Oncology, Copenhagen, Herlev, Denmark

REFERENCES:
- [Derived] Borch TH, Andersen R, Ellebaek E, Met O, Donia M, Svane IM. Future role for adoptive T-cell therapy in checkpoint inhibitor-resistant metastatic melanoma. J Immunother Cancer. 2020 Jul;8(2):e000668. doi: 10.1136/jitc-2020-000668. PMID 32747469

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was enrolled in the trial and started vemurafenib, but had rapid progression of a brain metastasis and it was deemed unsafe to continue with protocol treatment. Thus, the patient was excluded before receiving T cell infusion and did not complete treatment.
Groups:
- T Cell Therapy With Vemurafenib Pretreatment: 7 days before tumor harvest, patients will begin taking vemurafenib until admission for lymphodepleting chemotherapy followed by TIL infusion and interleukin-2.
  Vemurafenib: Patients will start treatment in a dose of 960 BID 7 days before tumor harvest and ends at the day of admission (day -8).
  Lymphodepleting chemotherapy regimen consisting of cyclophosphamide 60 mg/kg for 2 days and fludarabine 25 mg/m2 for 5 days (constitutes day -7 to -1 of admission).
  TIL infusion: A tumor is surgically removed in order to isolate, activate and expand tumor infiltrating lymphocytes (TIL) to high numbers. In vitro preparation usually takes 4-6 weeks using the young TIL method.
  On day 0 patients receive an infusion of TIL (1x10e9-2x10e11 cells).
  Interleukin-2 is administered according to the decrescendo regimen (18 MIU/m2 for 6 hours, 18 MIU/m2 for 12 hours, 18 MIU/m2 for 24 hours followed by 4,5 MIU/m2 for another 3 x 24 hours)
Period: Overall Study
Arm/Group | T Cell Therapy With Vemurafenib Pretreatment
Started | 13
Completed | 12
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | T Cell Therapy With Vemurafenib Pretreatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Stage at inclusion [Count of Participants; unit: Participants] — Staging according to the AJCC melanom staging 7th edition. M1a - Distant skin, subcutaneous, or nodal mets - and a normal serum LDH M1b - Lung metastases - and a normal serum LDH M1c - All other visceral metastases and a normal serum LDH OR any distant metastasis with an elevated serum LDH.
  Patients have progressively worse prognosis through the categories (M1a better -> M1c worse)
  Participants
    M1a | 1
    M1b | 1
    M1c | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Reported Adverse Events
Description: Determine the safety of the administration of vemurafenib in combination with TIL therapy including lymphodepleting chemotherapy and interleukin-2 treatment by collecting adverse events according to CTCAE v. 4.0. From start of treatment until 24 weeks after T cell infusion.
Time Frame: 0-40 weeks
Measure: Number; unit: Treatment related adverse events
Arm/Group | T Cell Therapy With Vemurafenib Pretreatment
Number analyzed (Participants) | 12
Treatment related adverse events
  Total | 124
  Grade 1-2 | 89
  Grade 3-4 | 35

2. Secondary Outcome: Treatment Related Immune Responses
Description: Number of patients whose infusion product contained anti-tumor reactive T cells by in vitro testing.
  Anti-tumor reactive T cells is defined by positive staining for two of the three markers (interferon gamma, tumor necrosis factor alpha and CD107a) in an intracellular cytokine staining using flow cytometry.
Time Frame: 0-24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Therapy With Vemurafenib Pretreatment
Number analyzed (Participants) | 12
Participants | 10

3. Secondary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1): Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Therapy With Vemurafenib Pretreatment
Number analyzed (Participants) | 12
Participants | 9

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS), defined as the time from the start of treatment to death, will be described with the Kaplan-Meier curve.
Time Frame: Up to 40 months
Measure: Median (Full Range); unit: Months
Arm/Group | T Cell Therapy With Vemurafenib Pretreatment
Number analyzed (Participants) | 12
Months | 28.8 [5.2 to 39.9]

5. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS), defined as the time from start of treatment to disease progression, relapse or death due to any cause, whichever is earlier, will be described with the Kaplan-Meier curve.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 40 months
Measure: Median (Full Range); unit: Months
Arm/Group | T Cell Therapy With Vemurafenib Pretreatment
Number analyzed (Participants) | 12
Months | 4.8 [2.5 to 36.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment until 24 weeks after T cell infusion.
Description: Adverse events were collected continually and as a minimum systematically at baseline, each treatment visit and at follow-up visits until 24 weeks after T cell infusion.
Arm/Group | T Cell Therapy With Vemurafenib Pretreatment
All-Cause Mortality (participants affected / at risk) | 7/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T Cell Therapy With Vemurafenib Pretreatment (N=12)
Pyrexia (General disorders) | 2 (2) — Pyrexia without neutropenia
Pancreatitis (Endocrine disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) — Colitis related to prior systemic anti-cancer treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T Cell Therapy With Vemurafenib Pretreatment (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (12)
Infection (Infections and infestations) | 5 (5)
Pyrexia (General disorders) | 1 (1) — Pyrexia without neutropenia
Fatique (General disorders) | 12 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Oral mucositis (Gastrointestinal disorders) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2)
Hallucination (Psychiatric disorders) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (13)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Rhinitis atrophic (Immune system disorders) | 1 (1)
Electrocardiogram QT prolonged (Cardiac disorders) | 3 (3)
Papilloma (Skin and subcutaneous tissue disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 5 (5)
Hepatic enzyme increased (Hepatobiliary disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 12 (13)
Lymphopenia (Blood and lymphatic system disorders) | 12 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT02354690/Prot_SAP_000.pdf